CLINICAL TRIAL: NCT00567359
Title: A Phase II Trial of Adjuvant Erlotinib in Patients With Resected, Early Stage Non-Small Cell Lung Cancer (NSCLC) With Confirmed Mutations in the Epidermal Growth Factor Receptor (EGFR)
Brief Title: Erlotinib in Patients With Resected, Early Stage NSCLC With Confirmed Mutations in the EGFR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Lecia V. Sequist, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-259
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; erlotinib; epidermal growth factor receptor; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Experimental)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Oral drug taken daily around the same time. Starting dose is 150mg once daily.
  Other Names: Tarceva

SUMMARY:
In this research study erlotinib will be given to eligible participants whose lung cancer has been removed by surgery. Eligible patients have adenocarcinoma, a type of non-small lung cancer, and must have 1 or more of the following characteristics: be female, be of Asian or Pacific Rim descent and/or be a never smoker. The potential participant's tumor will be examined for Epidermal growth factor (EGFR) mutations. EGFR is a protein that is overexpressed in most non-small cell lung cancers. Some EGFR has been found to have specific mutations and the participant must have one of these mutations in his tumor.

Erlotinib blocks this protein and may control tumor growth and increase survival. Previous research has shown that erlotinib is most effective for people who have these specific mutations in the EGFR.

DETAILED DESCRIPTION:
* Erlotinib is a pill taken daily and participants may continue to receive erlotinib for up to two years, as long as the cancer does not return and they do not experience any unacceptable side effects.
* While participants are receiving erlotinib, they will be asked to return to the clinic for study visits to monitor the status of their disease and their general health. For the first 5 months of erlotinib, they will return to the clinic monthly. After that they will return to the clinic every three months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of NSCLC of adenocarcinoma histology
* Stage IA-B, IIA-B, or IIIA by the American Joint Committee on Cancer 7th edition staging criteria
* Patients must have undergone surgical resection with curative intent within 6 months of enrollment
* Sufficient tumor tissue available for EGFR mutation analysis
* At least ONE of the following patient characteristics: previously detected deletion 19 or L858R EGFR mutation, female sex, history of never smoking, or Asian/Pacific Rim ethnicity (to be enrolled in the screening portion of trial).
* 18 years of age or older
* Tumor samples must have either exon 19 deletion mutations or the exon 21 L858R point mutation
* ECOG Performance status of 0,1, or 2
* Adequate organ function as outlined in protocol

Exclusion Criteria:

* Radiographic evidence of recurrent NSCLC prior to erlotinib treatment
* Confirmed T790M resistance mutation in the primary tumor sample
* Prior exposure to EGFR tyrosine kinase inhibitors
* Known hypersensitivity to erlotinib, gefitinib, or any closely related drug
* Pregnant or breastfeeding women
* Any evidence of clinically active interstitial lung disease
* Current use of enzyme-inducing anti-epileptic drugs, including carbamazepine, oxcarbazepine, phenytoin, fosphenytoin, phenobarbital, and primidone
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study
* Use of any non-FDA approved or investigational agent within 2 weeks of enrolling onto the trial, or failure to recover from the side effects of any of these agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lecia V. Sequist, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (8):
- United States (8):
  - Stanford University, Stanford, California
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - North Shore Medical Center, Peabody, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Taussig Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib
Started | 100
Completed | 99
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 100
Age, Continuous [Median (Full Range); unit: years] | 63 [41 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Asian | 83
  Asian | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100
Smoking Status [Count of Participants; unit: Participants]
  Never | 59
  <=10 pack years | 14
  >10 pack years + current | 27
Stage [Count of Participants; unit: Participants] — Cancer stage is a measure of disease progression. The later stage indicates more advanced cancer. So, the Participants with Stage II cancer have more advanced disease than stage I participants. The letters represent sub groups within a given stage, with B representing more advanced cancer than A.
  Participants
    Stage IA | 14
    Stage IB | 31
    Stage IIA | 11
    Stage IIB | 16
    Stage IIIA | 28
EGFR Mutation [Count of Participants; unit: Participants] — Epidermal Growth Factor Receptor (EGFR) allows healthy cells to grow and divide. A mutation in the EGFR gene can lead to cells having too many receptors. This can cause the cells to continue to grow and divide more than normal tissue, as happens in cancer.
  Participants
    Exon 19 Deletion | 62
    L858R | 35
    G719X | 2
    L861Q | 1

OUTCOME MEASURES:

1. Primary Outcome: 2-year Disease-free Survival
Description: The number of participants alive and free from disease recurrence 2 years after enrollment. Participants were monitored for disease recurrence with the use of surveillance radiographs. When possible and medically appropriate, tissue biopsies were obtained to prove recurrence.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 100
Participants | 88

2. Secondary Outcome: Number of Participants With Treat Related Serious Adverse Events
Description: Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE 3.0) from the start of treatment until 30 days after the end of treatment. Serious adverse events were defined as adverse events that were grade 3 or greater and deemed to be possibly, probably or definitely related to the study treatment.
Time Frame: From the start of treatment until 30 days after the end of treatment, up 13 months total
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 100
Participants | 20

3. Secondary Outcome: Median Overall Survival
Description: The median amount of time from the time of registration until death due to any cause
Time Frame: From the time of registration until death, up to approximately 9 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Erlotinib
Number analyzed (Participants) | 100
years | NA [NA to NA] — insufficient number of participants with events

4. Secondary Outcome: Median Disease Free Survival
Description: The median amount of time measured from the time of registration until the time of disease recurrence or death.
Time Frame: From registration to disease recurrence or death, up to approximately 9 years
Population: Median Disease Free Survival had not been met by the time of data cutoff.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Erlotinib
Number analyzed (Participants) | 100
years | NA [NA to NA] — insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment, up to 13 months total
Description: Further descriptions are not available for adverse events listed as 'Other' under an organ system.
Arm/Group | Erlotinib
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 20/100
Other Adverse Events (participants affected / at risk) | 99/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=100)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Hepatic-other (Hepatobiliary disorders) | 1 (1)
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 13 (15)
Skin-other (Skin and subcutaneous tissue disorders) | 1 (1)
Tearing (Eye disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=100)
Hemoglobin (Blood and lymphatic system disorders) | 5 (7)
Leukocytes (Investigations) | 5 (5)
Fatigue (General disorders) | 63 (92)
Dry skin (Skin and subcutaneous tissue disorders) | 49 (68)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (19)
Nail changes (Skin and subcutaneous tissue disorders) | 27 (40)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 24 (34)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 22 (38)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 74 (163)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 8 (11)
Skin-other (Skin and subcutaneous tissue disorders) | 26 (35)
Anorexia (Metabolism and nutrition disorders) | 13 (18)
Constipation (Gastrointestinal disorders) | 15 (22)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 74 (120)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 10 (14)
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 20 (31)
Nausea (Gastrointestinal disorders) | 31 (44)
Taste disturbance (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 11 (13)
GI-other (Gastrointestinal disorders) | 8 (11)
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 13 (15)
ALT, SGPT (Investigations) | 7 (7)
AST, SGOT (Investigations) | 7 (8)
Bilirubin (Investigations) | 8 (20)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 13 (13)
Anxiety (Psychiatric disorders) | 8 (9)
Neuropathy-sensory (Nervous system disorders) | 17 (21)
Dry eye syndrome (Eye disorders) | 13 (16)
Ocular-other (Eye disorders) | 13 (19)
Abdomen, pain (Gastrointestinal disorders) | 7 (7)
Back, pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Head/headache (Nervous system disorders) | 11 (14)
Joint, pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle, pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain-other (General disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (58)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 31 (48)
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 13 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-10-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT00567359/Prot_SAP_000.pdf